CLINICAL TRIAL: NCT02405533
Title: Phase II Randomized, Double-blind, Placebo-controlled Evaluation of AHCC (Active Hexose Correlated Compound) for the Eradication of HPV Infections in Women With HPV Positive Pap Smears
Brief Title: Phase II Evaluation of AHCC for the Eradication of HPV Infections
Acronym: AHCC4HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Judith A. Smith, Associate Professor & Director of WHIM Research Program, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-14-0866
Record Dates: First submitted 2015-03-17; First posted 2015-04-01 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Human Papilloma Virus; Dysplasia; CIN1; CIN2
Keywords: AHCC; nutritional supplement; HPV
MeSH Terms: interventions — Active Hexose Correlated Compound

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo control phase II study that patients receive either AHCC or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): AHCC 3 grams once a day on an empty stomach x 6 months then placebo once a day x 56 months.
  Interventions: Dietary Supplement: AHCC 3 grams once a day
- Group 2 (Placebo Comparator): Placebo once a day on an empty stomach x 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AHCC 3 grams once a day — AHCC supplementation x 6 months with Placebo x 6 months
  Other Names: active hexose correlated compound
  Arms: Group 1
Other: Placebo — Placebo supplementation x 12 months
  Arms: Group 2

SUMMARY:
This is a phase II randomized, double-blind placebo-controlled, crossover trial. The primary outcome of this trial is achieving durable eradication persistent high risk HPV infection determined by HPV negative test results achieved while on active treatment with AHCC and maintained for 6 month post supplementation and 12 months post completion of AHCC treatment compared to placebo.

DETAILED DESCRIPTION:
This is a phase II randomized, double-blind placebo-controlled, crossover trial. The primary outcome of this trial is achieving durable eradication HPV infection determined by HPV negative test results achieved while on active treatment with AHCC and maintained for 6 month post supplementation and 12 months post completion of AHCC treatment for Group 1. We will follow all patients for at least 12 months and up to 30 months depending on success of achieving a negative HPV testing results. After receiving AHCC 3 grams x 6 months if positive at the end of 12 months of study treatment, they are considered a treatment failure. If negative after completion of 6 months of AHCC supplementation + 6 months of placebo, they will continue on study for another six months (2 visits) to confirm they remain HPV negative and durable response. Group 2 will serve as untreated control for all time points (end of supplementation, then 6, 9, and 12 months post end of AHCC supplementation.

ELIGIBILITY:
Inclusion Criteria:

* • Women over 30 years of age who have a HPV positive test and normal/negative cytology, atypical cells, ASCUS, or CIN1 or CIN2 cervical dysplasia within three months of study entry.

  * Women must have had 2 other HPV positive tests with normal/negative cytology, atypical cells, ASCUS, or CIN1 or CIN2 cervical dysplasia

    * 1 greater than 6 months and no more than 18 months prior to study entry
    * 1 greater than 24 months prior to study entry.
  * Women of child bearing potential must have a negative urine pregnancy test within 7 days of therapy start.
  * Patients must have adequate hematologic, renal, and hepatic function as noted from labs within the previous 12 months: ANC >/= 1,500 cells/mm3, platelets 100,000 >/= cells/mm3; Creatinine clearance>/= 60 mL/min (estimated by Cockcroft Gault equation), total bilirubin, SGPT, SGOT, and alkaline phosphatase </= 1.5 times normal.
  * Patients of child-bearing age must agree to use effective methods of contraception (oral contraceptives, condoms, etc.) while on study.

Exclusion Criteria:

* • History of myocardial infarction within past 6 months, unstable angina, CHF, or uncontrolled hypertension (> 140/90).

  * Women with a current or prior diagnosis of cancer
  * Women with a current diagnosis of CIN3 cervical dysplasia
  * Women that are pregnant or breast feeding.
  * Women with a history of Hepatitis (autoimmune, A, B, or C) or antigen positive
  * Patients with history of significant psychiatric disorders (schizophrenia, bipolar, psychosis) or uncontrolled seizures.
  * Patients with significant medical co-morbidities at the discretion of the primary Gynecologist. Including immunosuppressive conditions (i.e. HIV+, rheumatoid arthritis, etc) or taking immune modulation mediations (i.e. immunosuppressants)
  * Women that have taken AHCC within the past six months.
  * Women currently taking other immune modulating nutritional supplements.
  * Patients who have undergone a hysterectomy (supracervical hysterectomy allowed)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Roche, COBAS HPV DNA Assay (Pleasanton, CA) | once every 3 months for 12 months up to 18 months
  HPV DNA testing

SECONDARY OUTCOMES:
Interferon beta | once every 3 months for 12 months up to 18 months
  Evaluation of Interferon Beta level
Interferon gamma | once every 3 months for 12 months up to 18 months
  Evaluation of Interferon gamma level
NK Cells | once every 3 months for 12 months up to 18 months
  Evaluation of Natural Killer (NK) cells

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Smith, Pharm.D., Study Chair — UTTexas_Houston
Locations (1):
- UTHealth Medical School at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Smith JA, Gaikwad AA, Mathew L, Rech B, Faro JP, Lucci JA 3rd, Bai Y, Olsen RJ, Byrd TT. AHCC(R) Supplementation to Support Immune Function to Clear Persistent Human Papillomavirus Infections. Front Oncol. 2022 Jun 22;12:881902. doi: 10.3389/fonc.2022.881902. eCollection 2022. PMID 35814366